CLINICAL TRIAL: NCT04783428
Title: Tumor-induced Osteomalacia Disease Monitoring Program (TIO DMP)
Brief Title: Tumor-induced Osteomalacia Disease Monitoring Program
Status: Active, not recruiting | Type: Observational
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: UX023T-CL403
Record Dates: First submitted 2021-02-18; First posted 2021-03-05 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Tumor-induced Osteomalacia (TIO)
MeSH Terms: conditions — Oncogenic osteomalacia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Prior TIO Burosumab Clinical Trial Participants
  Interventions: Other: No intervention
- Adults Who Have Not Participated In Prior Burosumab Clinical Trials
  Interventions: Other: No intervention
- Pediatrics Who Have Not Participated In Prior Burosumab Clinical Trials
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Access to any treatment is through authorized commercial use and not as part of this DMP

SUMMARY:
The objectives of this observational study are to assess the long-term safety and long-term effectiveness of burosumab in patients with TIO who are being treated with burosumab as prescribed by their physician and to monitor the course of the underlying phosphaturic mesenchymal tumor (PMT) overtime in patients with TIO irrespective of their treatment status.

DETAILED DESCRIPTION:
Enrolled patients may or may not be treated with commercially available burosumab during the TIO DMP at the discretion of their treating physician. Given the observational nature of the TIO DMP, specific treatments or supportive management will not be provided as part of the study.

ELIGIBILITY:
Inclusion Criteria:

* Have a clinical diagnosis of TIO based on the presence of an underlying PMT (confirmed by imaging) AND/OR historical documentation. Note: For adult patients with TIO in whom the causative PMT has never been located, and all pediatric patients, documented evidence of negative genetic testing for other hereditary hypophosphatemic disorders is necessary
* For patient safety, all participating female patients of child-bearing potential must be willing to have pregnancy tests prior to certain assessments performed as part of the DMP
* Be willing to provide access to prior medical records including tumor pathology reports and biopsy slides, imaging, biochemical, and diagnostic, medical, and surgical history data, if available
* Be willing and able to provide informed consent after the nature of the study has been explained, and prior to any research-related procedures
* Be willing and able to comply with the study visit schedule and study procedures

Exclusion Criteria:

* Have a clinical diagnosis of TIO deemed to be caused by a tumor other than a PMT
* Serious medical or psychiatric comorbidity that, in the opinion of the Investigator, would present a concern for patient safety or compromise the ability to provide consent or comply with the study visit schedule and study procedures
* Less than 1 year of life expectancy (for any cause) in the opinion of the Investigator
* Concurrent enrollment in a clinical trial without prior approval from the TIO DMP Sponsor
* Undergoing treatment with burosumab for an unapproved indication

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: May include patients who have undergone complete tumor resection and continue to have biochemical/clinical evidence of disease, patients with tumor identified, or patients in whom causative tumor has not been identified and who have been diagnosed with TIO based on biochemical/clinical symptom profile.
  Patients may be treated with burosumab, or phosphate and active vitamin D metabolites/analogs, as prescribed by a physician, or may be untreated, at any time during the TIO DMP.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2032-02-28 (Estimated); Study Completion 2032-02-28 (Estimated)

PRIMARY OUTCOMES:
Long-Term Effectiveness of Burosumab: Change From Baseline in Serum Phosporus Over Time | 10 years
Long-Term Effectiveness of Burosumab: Change From Baseline in Serum 1,25(OH)2D Over Time | 10 years
Long-Term Effectiveness of Burosumab: Change From Baseline in Serum Alkaline Phosphatase (ALP) Over Time | 10 years
Long-Term Effectiveness of Burosumab: Change From Baseline in Serum FGF23 Over Time in Participants Not Undergoing Treatment With Burosumab | 10 years
Long-Term Safety of Burosumab: Change From Baseline in Phosphaturic Mesenchymal Tumor (PMT) Size Over Time as Assessed by Tumor Imaging | 10 years
Long-Term Safety of Burosumab: Number of Participants With New PMT Development as Assessed by Tumor Imaging | 10 years
Long-Term Safety of Burosumab: Change From Baseline in Serum iPTH Over Time | 10 years
Long-Term Safety of Burosumab: Change From Baseline in Serum Calcium Over Time | 10 years
Long-Term Safety of Burosumab: Change From Baseline in Urine Calcium Over Time | 10 years
Long-Term Safety of Burosumab: Change From Baseline Urinary Calcium/Creatinine Ratio | 10 years
Long-Term Safety of Burosumab: Change From Baseline in Serum Creatinine Over Time | 10 years
Long-Term Safety of Burosumab: Change From Baseline in Urine Creatinine Over Time | 10 years
Long-Term Safety of Burosumab: Change From Baseline in Urine Protein/Creatinine Ratio Over Time | 10 years
Long-Term Safety of Burosumab: Number of Participants With Nephrocalcinosis Over Time | 10 years
Long-Term Safety of Burosumab: Number of Participants With Serious Adverse Events (SAEs) and Adverse Events (AEs) and Related AEs | 10 years
Long-Term Safety of Burosumab: Number of Participants With Incidence and/or Progression of Spinal Stenosis Over Time | 10 years
Long-Term Safety of Burosumab: Number of Participants With Normal and/or Potentially Clinically Significant Pregnancy Outcomes | 10 years
  Includes maternal, neonatal and infant outcomes
Long-Term Effectiveness of Burosumab: Change From Baseline in Brief Fatigue Inventory (BFI) Scores in Adult Participants Over Time | 10 years
Long-Term Effectiveness of Burosumab: Change From Baseline in Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue Scores in Pediatric Participants Over Time | 10 years
Long-Term Effectiveness of Burosumab: Change From Baseline in Brief Pain Inventory (BPI) Scores in Adult Participants Over Time | 10 years
Long-Term Effectiveness of Burosumab: Change From Baseline in PROMIS Pain Scores in Pediatric Participants Over Time | 10 years
Long-Term Effectiveness of Burosumab: Change From Baseline in PROMIS Physical Function Scores Over Time | 10 years
Long-Term Effectiveness of Burosumab: Change From Baseline in Short Form-36 version 2 (SF-36v2) in Adult Participants Over Time | 10 years
Long-Term Effectiveness of Burosumab: Change in Short Form-10 (SF-10) for Pediatric Participants Over Time | 10 years
Long-Term Effectiveness of Burosumab: Number of Participants With Changes From Baseline in Clinical Findings | 10 years
Long-Term Effectiveness of Burosumab: Number of Participants With Changes From Baseline in Resource/Health Utilization | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Ultragenyx Pharmaceutical Inc
Locations (6):
- United States (5):
  - Yale University, New Haven, Connecticut
  - Indiana University, Bloomington, Indiana
  - Johns Hopkins University, Baltimore, Maryland
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Virginia, Charlottesville, Virginia
- IDIM - Instituto de Diagnóstico e Investigaciones Metabólicas, Buenos Aires, Argentina

REFERENCES:
- See also: Ultragenyx Patient Advocacy/TIO Disease Information — https://ultrarareadvocacy.com/tumor-induced-osteomalacia-tio/
- See also: Ultragenyx Transparency Commitment — http://www.ultragenyx.com/our-research/our-clinical-trial-transparency-commitment/